CLINICAL TRIAL: NCT02184962
Title: "Levels of RANKL and OPG in Gingival Crevicular Fluid of Patients With Post-menopausal Osteoporosis / Osteopenia and Periodontal Disease."
Brief Title: Periodontal Disease and Post-menopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Córdoba (Other)
Responsible Party: Principal Investigator, María Eugenia Verde, María Eugenia Verde - Cátedra de Periodoncia A - UNC, Universidad Nacional de Córdoba
Other Study IDs: MEV-2030; UNC-2013 (Registry Identifier: UCordoba)
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Osteoporosis; Osteopenia; Periodontal Disease
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study was to investigate the levels of RANKL and Osteoprotegerin, and their relationship in gingival crevicular fluid of post-menopausal women with osteoporosis/osteopenia and chronic periodontitis simultaneously and evaluate the effect that the use of bisphosphonates in periodontal disease.

Study hypothesis:

"The osteoporosis / osteopenia in postmenopausal women patients with periodontal disease affect the ratio RANKL / OPG in gingival crevicular fluid samples favoring osteoclastogenesis processes "

DETAILED DESCRIPTION:
81 active periodontal sites from 31 postmenopausal women aged 45-70 years with chronic periodontitis were studied. Samples of gingival crevicular fluid were collected by paper strips and ELISA test was conducted to determine the total concentration of RANKL, OPG, and then obtain the values of the RANKL / OPG ratio. We analyzed 66 samples of gingival crevicular fluid obtained from active periodontal sites of 17 patients with osteopenia / osteoporosis and 15 samples gingival crevicular fluid obtained from active periodontal sites obtained of 14 controls patients with normal osseous condition.

Statistical analyzes were computed and analyzed using Graphpad Software. To determine if the data correspond to a normal distribution the D'Agostino-Pearson test was used. The values of cytokines (RANKL and OPG) and its ratio (RANKL / OPG) were compared using Mann-Whitney Test t U. Analysis Spearman correlation and linear regression for statistic was also performed to determine whether there was any relationship between the variables analyzed. It was considered as statistically significant p value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45-70 years with Absorptiometry Dual Energy X-ray (DEXA).

  * Control group: post-menopausal women with periodontal disease and normal osseous condition.
  * Study group: post-menopausal womens with periodontal disease and osteoporosis/osteopenia with and without bisphosphonate treatment (risedronate or ibandronate 150 mg) for longer than 3 months before the study and another.

Exclusion Criteria:

* Patients with history of aggressive periodontitis and had received any periodontal treatment when they entered the study
* Patients with any systemic illness (except osteopenia/osteoporosis)
* Patients who received antibiotic or non-steroidal anti-inflammatory therapy in the 6 months prior to the study.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteopenia / osteoporosis and controls with normal osseous condition. Both groups with chronic periodontitis
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
levels of RANKL and OPG | one year

CONTACTS AND LOCATIONS:
Overall Officials: María E Verde, Odontóloga, Principal Investigator — Facultad de Odontología - UNC
Locations (1):
- Facultad de Odontología - Universidad Nacional de Córdoba, Córdoba, Córdoba Province, Argentina